CLINICAL TRIAL: NCT02527980
Title: E-Cigarettes: Dynamic Patterns of Use and Health Effects
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2015-0575; A534252 (Other: UW Madison); SMPH\MEDICINE\TOBACCO RE (Other: UW Madison); 1R01CA190025-01 (NIH)
Record Dates: First submitted 2015-08-14; First posted 2015-08-19 (Estimated); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Smoking; Nicotine Dependence
Keywords: electronic cigarettes; nicotine dependence; smoking; tobacco use
MeSH Terms: conditions — Smoking; Tobacco Use Disorder; Vaping; Tobacco Use

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine samples retained for additional analyses
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- dual users: Individuals who at the point of study enrollment are using both electronic cigarettes (ecig) and commercial cigarettes (CCs)
  Interventions: Other: No intervention: observation only
- commercial cigarette (CC) only users: Individuals who at the point of study enrollment are using exclusively commercial cigarettes
  Interventions: Other: No intervention: observation only

INTERVENTIONS:
Other: No intervention: observation only — For all participants: We will conduct a 2-year longitudinal cohort study comprising participants who smoke exclusively CCs (n=175) and dual users of e-cigs and CCs (n=275). We will use state-of-the-art ecological momentary assessments to determine: 1) dynamic patterns of e-cig and CC use and related outcomes (e.g., dependence, withdrawal symptoms, CC quit attempts and quitting success); 2) episodic (affective, contextual, social) and stable person-factor (lifestyle factors, demographics) variables that covary meaningfully with e-cig and CC use and related outcomes; and 3) biomarkers of tobacco and carcinogen exposure as well as other health-related outcomes (e.g., reduced pulmonary function.

SUMMARY:
The proposed research will provide in-depth, longitudinal data, based on real-time reports, which will address key priorities for the FDA including, increased understanding of the relations between electronic cigarette (e-cig) use and 1) nicotine dependence, 2) reductions in combustible cigarette (CC) use, 3) attempts to quit CC use and the success of those attempts, and 4) health-related outcomes such as biomarkers of exposure and carcinogenicity.

DETAILED DESCRIPTION:
Primary Aim: Characterize e-cig use patterns both acutely and over 2 years and relate them to patterns of CC use (including reduced CC use), nicotine dependence and related variables (e.g., withdrawal suppression), and attempts and success in quitting CC use. Investigators will use ecological momentary assessment (EMA) to obtain fine grained, real-time data on e-cig and CC use. These data will be used to test the hypotheses that increasing and higher levels of e-cig use, measured in real-time, will be negatively related to CC use, nicotine dependence, and CC withdrawal severity and positively related to CC quit attempts and CC cessation success.

Secondary Aim 1: Determine how the use of e-cigs is related to biomarkers of tobacco exposure and cancer risk, and to acute and chronic pulmonary health outcomes. Investigators will examine the relation between e-cig use and cancer biomarkers, exposure biomarkers, and pulmonary function.

Secondary Aim 2: Identify person factors, contextual variables, and patterns of behaviors and symp-toms that predict e-cig and CC use patterns and key outcomes (e.g., CC cessation, health-related outcomes), and identify variables that moderate relations between e-cig use and such outcomes. Investigators will attempt to identify contextual variables and person factors that predict increased e-cig use, decreased CC use (including cessation), reduced nicotine dependence, and significant changes in biomarkers and health outcomes. Further, investigators will identify variables that moderate such relations, revealing factors and events that make changes in e-cig and CC use, and associated outcomes, especially likely.

ELIGIBILITY:
Inclusion Criteria:

* Specific eligibility requirements are:

  1. ≥ 18 years old
  2. able to read and write English
  3. no plans to quit smoking and/or e-cig use in the next 30 days
  4. not currently taking smoking cessation medication
  5. not currently in treatment for psychosis or bipolar disorder
  6. participants must report either that they have:
* smoked at least 5 cigarettes per day for the past 6 months and not used e-cigs within the last 3 months ("exclusive smokers")
* used nicotine-containing e-cigs at least once a week for the past month and have smoked at least 5 CCs/day for the last 3 months ("dual users").

Exclusion Criteria:

* Individuals not meeting any one of the inclusion criteria. Those not meeting any one (or more) of criteria 1-5 and either criterion 6a or 6b will be excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 2 groups: regular users of electronic cigarettes and commercial cigarettes and regular exclusive users of commercial cigarettes
Sampling Method: Non-Probability Sample
Enrollment: 422 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Characterize patterns of ecig and CC use | 2 years
  To address the primary aim of understanding dynamic use patterns in an observational cohort, investigators will assess the use of CCs, e-cigs and other tobacco use-related behavior. E-cig attitudinal questions and questions about e-cig use in the environment will be asked. Investigators will assess person factors that may inform understanding of who is using e-cigs and in what manner these may also moderate the effects of e-cig use. Investigators will also use ecological momentary assessment (EMA) to obtain data on e-cig and CC use. Investigators will assess exhaled carbon dioxide, cotinine and polycyclic aromatic hydrocarbons (PAHs). Pulmonary function will be assessed via spirometry conducted in accordance with the American Thoracic Society guidelines. Investigators will also assess prior pulmonary diagnoses. Participants will also complete the St. George Respiratory Questionnaire for chronic obstructive pulmonary disease (SGRQ-C).

CONTACTS AND LOCATIONS:
Overall Officials: Megan E Piper, Phd, Principal Investigator — UW-CTRI
Locations (2):
- United States (2):
  - CTRI Monroe, Madison, Wisconsin
  - CTRI Milwaukee, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Piper ME, Baker TB, Benowitz NL, Jorenby DE. Changes in Use Patterns Over 1 Year Among Smokers and Dual Users of Combustible and Electronic Cigarettes. Nicotine Tob Res. 2020 Apr 21;22(5):672-680. doi: 10.1093/ntr/ntz065. PMID 31058284